CLINICAL TRIAL: NCT02822586
Title: Phase 1B Trial: Evaluation of the Safety of Adding Brentuximab Vedotin to Low-Dose Total Skin Electron Beam (TSEB) for Treatment of Patients With Mycosis Fungoides and Sézary Syndrome
Brief Title: TSEB and Brentuximab for Treatment of Mycosis Fungoides & Sezary Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15-10917; IST2015100830 (Other: Seattle Genetics); NCI-2016-01509 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Mycosis Fungoides; Sézary Syndrome
Keywords: CD30-positive; Stage IB to Stage IVA
MeSH Terms: conditions — Mycosis Fungoides; Sezary Syndrome | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Stage IB and Stage IIA to IIIB [if N0-1]) (Experimental): (Eligible patients with Stage IB, IIA, IIB, and IIIA [if N0-1])
  Brentuximab Vedotin 1.8 mg/kg IV every 3 weeks for 3 doses beginning 3 weeks prior to initiation of TSEB.
  TSEB 12 Gy in 6 fractions at 2 Gy/fraction treated twice/week.
  Interventions: Radiation: TSEB Therapy; Drug: Brentuximab vedotin
- Cohort B(Stage IIA to IIIB; IVA;transformed CTCL) (Experimental): (Eligible patients with Stage IIA, IIB, IIIA [if N2-3]; IIIB; Stage IVA; and transformed CTCL)
  Brentuximab Vedotin 1.8 mg/kg IV every 3 weeks for 3 doses beginning 3 weeks prior to initiation of TSEB.
  TSEB 12 Gy in 6 fractions at 2 Gy/fraction treated twice/week.
  Continuation of brentuximab every 3 weeks until disease progression or unacceptable toxicity or for up to 2 years as a study participant, (whichever occurs first).
  Interventions: Radiation: TSEB Therapy; Drug: Brentuximab vedotin

INTERVENTIONS:
Radiation: TSEB Therapy — TSEB is a type of radiation treatment in which the skin over the whole body is treated with electron radiation beams. All participants will receive the same standard TSEB dose and treatment schedule. During TSEB, patients are treated in a standing position on a rotating platform.
  Other Names: total skin electron beam; TSEB
Drug: Brentuximab vedotin — An antibody-drug conjugate (ADC) that targets CD30. A standard dose of brentuximab vedotin will be administered to all patients by intravenous infusion 3 weeks prior to initiation of TSEB and then every 3 weeks for 3 cycles.
  Other Names: Adcetris

SUMMARY:
The purpose of this study is to evaluate the cutaneous toxicity and treatment response associated with administering concurrent TSEB and brentuximab vedotin in patients with mycosis fungoides or Sézary Syndrome.

DETAILED DESCRIPTION:
This study is a 2-cohort, open-label, phase 1B trial to evaluate the cutaneous toxicity, overall toxicity, and treatment response associated with administering concurrent low-dose TSEB and brentuximab vedotin in patients with mycosis fungoides or Sézary Syndrome. Duration of complete skin response, DOCB, and tumor response in lymph nodes and blood will also be evaluated. Additionally, skin-related QOL and neurotoxicity will be assessed.

Patients will be enrolled in 1 of 2 cohorts based on disease stage.

Cohort A will include patients with earlier stage disease (selected Stage IB in patients who have had one previous course of therapy) and Stages IIA through IIIA [if N0-1]).

Cohort B will include patients with more advanced disease (Stage IIA through IIIA [if N2-3], Stage IIIB, Stage IVA, and transformed CTCL) who are candidates for low-dose TSEB and/or systemic therapy.

A standard dose of brentuximab vedotin will be administered to all patients by intravenous infusion 3 weeks prior to initiation of low-dose TSEB and then every 3 weeks for a total of 3 cycles. Cohort A patients will complete brentuximab vedotin after 3 cycles; patients in Cohort B will continue brentuximab vedotin until disease progression or unacceptable toxicity, whichever occurs first. In the absence of progression or unacceptable toxicity, the patient may receive brentuximab vedotin for up to 2 years as a study participant. A total of 12 Gy TSEB (ie, low-dose TSEB) will be administered to both cohorts per standard protocol in 6 fractions (2 fractions per week) beginning 3 weeks after the first dose of brentuximab vedotin.

The Modified Severity Weighted Assessment Tool (mSWAT) (16), completed by the investigator, will be used to determine skin involvement at baseline and skin response to treatment beginning after administration of the 3 doses of brentuximab vedotin and low-dose TSEB. Skindex-16, a patient-completed form that measures symptoms and perceptions of toxicity in patients with skin disease will be used to assess skin-related QOL. Additionally, Form NTX will be completed by patients in Cohort A to assess symptoms of CIPN which is a side effect of brentuximab vedotin.

The sample size for this study will be a maximum of 15 patients for a total of 12 evaluable patients with no more than 6 patients in Cohort B. However, if the number of patients with severe toxicity exceeds the established acceptable incidence, accrual will end before reaching the sample size goal of 12 evaluable patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CD30-positive (defined in this study as ≥ 1% expression) Mycosis Fungoides (including large cell transformation variant) or Sezary Syndrome who have either:

  * Received prior systemic therapy (for whom commercial supply of brentuximab vedotin is available) OR
  * Not received prior systemic therapy (who will receive brentuximab vedotin free of charge)
* Any of the disease stages listed below

  * Stage IB disease that meets one of the following criteria:
  * Plaque disease (ie,T2b staging)
  * Diffuse skin involvement with indication for TSEB (plaque disease with or without patches)
  * Not appropriate for treatment with focal therapies
  * One prior course of low-dose TSEB or one prior course of systemic chemotherapy regimens (excluding brentuximab)
  * Stage IIA, IIB, or IIIA that meets ONE or BOTH of the following criteria:
  * Patient is a candidate for treatment with low-dose TSEB
  * Patient is a candidate for systemic therapy
  * IIIB or IVA disease requiring systemic therapy
  * Transformed CTCL
* Candidate for TSEB based on investigator determination
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, 2, or 3, if the performance status of 3 is due to skin disease involvement
* Adequate bone marrow function as defined below:

  * Absolute neutrophil count (ANC) ≥ 1000/mm3
  * Platelets > 75,000/mm3
  * Hemoglobin ≥ 9 g/dL

    * Note: Patients requiring transfusion to meet the hemoglobin requirement are not eligible for the study.
* Calculated creatinine clearance (CrCl) > 30 mL/min.
* Adequate hepatic function as defined below:

  * Total bilirubin ≤ 1.5 x ULN for the laboratory
  * Aspartate aminotransferase (AST) ≤ 2 x ULN for the laboratory
  * Alanine aminotransferase (ALT) ≤ 2 x ULN for the laboratory
  * Prothrombin time with INR ≤ ULN for the laboratory
* A woman of childbearing potential (WCBP), defined as a woman who is < 60 years of age and has not had a hysterectomy, must have a documented negative serum pregnancy test 14 days prior to study registration

  * Note: If study treatment is not initiated within 7 days after the pregnancy test, the pregnancy test must be repeated.
* A WCBP and a male patient with a partner who is a WCBP must agree to use a medically accepted method for preventing pregnancy for the duration of study treatment and for at least 6 months following completion of study treatment
* Ability to understand and willingness to sign the consent form

Exclusion Criteria:

* Previous TSEB therapy with total dose > 20 Gy
* Previous brentuximab treatment
* Any of the following within 4-3 weeks prior to initiating study treatment

  * Systemic biologic therapy
  * Monoclonal antibody
  * Chemotherapy
  * TSEB
  * Phototherapy
  * Other investigational therapy
* Anticancer topical therapy, including therapeutic doses of steroids, within 2 weeks prior to initiating study treatment

  * Note: Topical steroids at doses intended for symptom management are permitted prior to study enrollment and may continue during study treatment.
* Peripheral sensory neuropathy or peripheral motor neuropathy ≥ grade 2 per NCI CTCAE v4.0
* Diabetic neuropathy (any grade)
* Demyelinating form of Charcot-Marie-Tooth Syndrome
* History of progressive multifocal leukoencephalopathy
* Active or clinically significant cardiac disease including any of the following:

  * Unstable angina (eg, anginal symptoms at rest) or onset of angina within 3 months prior to initiating study treatment
  * Myocardial infarction within 6 months prior to initiating study treatment
  * New York Heart Association (NYHA) class III or IV congestive heart failure (Appendix 4)
* Active ≥ grade 3 (per NCI CTCAE v4) viral, bacterial, or fungal infection within 2 weeks prior to initiation of study treatment
* Known human immunodeficiency virus (HIV) infection
* Known or suspected active hepatitis B or C infection
* Known cirrhosis
* Known Gilbert's Syndrome
* Planned ongoing treatment with another drug that may potentially have adverse interactions with brentuximab vedotin; if such a drug has been used, it must be discontinued at least 1 week prior to initiating study treatment (see Section 6.6); examples of potential interactions include:

  * Coadministration of strong inhibitors of CYP3A4 (eg, ketoconazole, ritonavir, clarithromycin)
  * Coadministration of CYP3A4 inducers (eg, rifampin)
  * Concomitant treatment with strong inhibitors of P-glycoprotein (P-gp)
* Known hypersensitivity to any excipient contained in the brentuximab formulation
* Prior malignancy or myelodysplastic syndrome (active within 3 years of screening) except completely excised non-invasive basal cell or squamous cell carcinoma of the skin, and in situ squamous cell carcinoma of the cervix
* Pregnancy or breastfeeding
* Medical, psychological, or social condition that, in the opinion of the investigator, may increase the patient's risk or limit the patient's adherence with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-04-29 (Actual)

PRIMARY OUTCOMES:
Cutaneous toxicity of combining TSEB and brentuximab vedotin in patients with MF or SS (Cohorts A and B). | 6 months
  Selected cutaneous adverse events (AEs) that occurred during treatment or during the 3 months following initiation of study treatment and that are characterized and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (NCI CTCAE v4.0) including ≥ grade 3 AEs and selected grade 2 AEs
Number of patients who achieved Complete Response (CR) and Partial Response(PR) | 2 years
  Number of patients who have achieved cutaneous CR to treatment defined as 100% clearance of skin lesions or cutaneous partial response (PR) defined as 50%-99% clearance of skin disease from baseline without new tumors in patients with T1-, T2-, or T4-only skin disease.

SECONDARY OUTCOMES:
Duration of complete skin response (Cohorts A and B) | 2 years
  Duration of skin response defined as the time from first determination of CR until relapse in the skin based on mSWAT assessment.
Tumor response in lymph nodes (Cohort B) | 6 months
  Tumor response in lymph nodes for patients with N2 or N3 disease at baseline.
Tumor response in blood (Cohort B) | 6 months
  Tumor response in blood for patients with B1 or B2 disease at baseline.
Overall Toxicity (Cohorts A and B) | 2 years
  AEs reported using criteria in the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE v4.0) and AEs defined in the protocol.
Skin-related Quality of Life (QOL) (Cohorts A and B) | 2 years
  Patient responses to questions on Skindex-16 (standardized assessment measures for patients with skin disease) that will be administered at baseline and at 2, 4, 10, and 16 weeks following completion of TSEB
Patient-reported chemotherapy-induced peripheral neuropathy (CIPN) (Cohort A) | 2 years
  Patient responses to questions on Form NTX (standardized patient-completed assessment tool to evaluate CIPN) that will be administered at baseline and at 2, 4, 10, and 16 weeks following completion of TSEB.
Duration of clinical benefit (DOCB) | 2 years
  DOCB defined as the time from initial response until any total skin-equivalent treatment (eg, topical treatment to > 50% of body surface, phototherapy, second TSEB treatment) or systemic therapy is initiated, or until disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Shiyu Song, M.D., Ph.D., Principal Investigator — Massey Cancer Center
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States